CLINICAL TRIAL: NCT00004480
Title: Study of Botulinum Toxin in Patients With Primary Hyperhidrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/14182; MTS-GCO-98-913NE; ALLERGAN-MTS-GCO-98-913NE
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-07

CONDITIONS: Hyperhidrosis
Keywords: dermatologic disorders; hyperhidrosis; rare disease
MeSH Terms: conditions — Hyperhidrosis; Skin Diseases; Rare Diseases | interventions — Botulinum Toxins, Type A

INTERVENTIONS:
Drug: botulinum toxin type A

SUMMARY:
OBJECTIVES:

I. Determine the optimal dose of botulinum toxin necessary to decrease sweating in patients with primary hyperhidrosis.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Patients receive injections of botulinum toxin in the clinical trial for 6 months. Patients undergo an iodine starch test and a sympathetic skin response test to assess the efficacy of the drug. Patients also complete questionnaires to evaluate the amount of sweating.

ELIGIBILITY:
* Diagnosis of hyperhidrosis
* Excessive sweating in the hands, feet, armpits, forehead, or body

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-07

CONTACTS AND LOCATIONS:
Overall Officials: Horacio Kaufmann, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States